CLINICAL TRIAL: NCT04217772
Title: Optical Coherence Tomography Angiography Analysis After Childhood Lensectomy
Brief Title: OCTA Analysis In Children After Lensectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Director of Cataract Department, Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OCTA-LZL
Record Dates: First submitted 2019-12-29; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Deprivation Amblyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eyes post-lensectomy (Experimental): Eyes of children after cataract surgery
  Interventions: Device: Optical Coherence Tomography Angiography
- Healthy Eyes (No Intervention): Eyes of healthy volunteers

INTERVENTIONS:
Device: Optical Coherence Tomography Angiography — A device testing the vascular density in the retina
  Arms: Eyes post-lensectomy

SUMMARY:
The aim of this study is to quantify and compare the foveal avascular zone (FAZ), the parafoveal and foveal vessel density of superficial (SCP) and deep capillary plexus (DCP) and retinal thickness in deprivation amblyopic eyes, fellow non-amblyopic eyes, and age-matched normal eyes, using optical coherence tomography angiography (OCTA). The FAZ, parafoveal and foveal SCP and DCP, and retinal thickness were measured in normal controls and at least 3 months postoperatively in children with unilateral cataract and compared between groups after adjusting for axial length and spherical equivalents.

ELIGIBILITY:
Inclusion Criteria:

* children after cataract surgery and healthy volunteers

Exclusion Criteria:

* presence of corneal opacity preventing detailed imaging
* nystagmus
* retinal disease,
* persistent fetal vasculature
* intraocular inflammation,
* glaucoma
* vitreoretinal surgery
* premature birth
* neurologic disease
* systemic disease that could alter microvasculature (including diabetes, hypertension, cardiovascular disease and renal disease)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Foveal retinal thickness | up to 36 months
  Foveal retinal thickness in microns
Area of foveal avascular zone | up to 36 months
  Area of foveal avascular zone in square microns

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, MD, Principal Investigator — Eye Hospital of WMU
Locations (2):
- China (2):
  - Eye Hospital of WMU, Hangzhou, Zhejiang
  - The affiliated Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No